CLINICAL TRIAL: NCT04003363
Title: The UK National Registry for Myotonic Dystrophy
Brief Title: The United Kingdom National Registry for Myotonic Dystrophy
Status: Recruiting | Type: Observational
Sponsor: Newcastle University (Other)
Responsible Party: Sponsor
Other Study IDs: 18/NE/0289
Record Dates: First submitted 2019-06-25; First posted 2019-07-01 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2022-11

CONDITIONS: Myotonic Dystrophy
Keywords: Myotonic Dystrophy; Myotonic Dystrophy Type 1; Myotonic Dystrophy Type 2; DM; DM1; DM2
MeSH Terms: conditions — Myotonic Dystrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with Myotonic Dystrophy
  Interventions: Other: Patient Registry

INTERVENTIONS:
Other: Patient Registry — Participants who have volunteered to participate will complete various questionnaires relating to their condition.

SUMMARY:
Myotonic dystrophy (dystrophia myotonica - DM) exists in two forms, usually referred to as DM1 (type 1) and DM2 (type 2). Both conditions are genetic disorders but each affects a different gene. DM1 is the most common adult-onset muscular dystrophy, and is thought to affect at least 1 in 8,000 people worldwide.

The aim is to facilitate a questionnaire based research study in order to better characterise and understand the disease in the UK. By maintaining a national registry this will help identify potential participants eligible for clinical trials in the future.

DETAILED DESCRIPTION:
The UK DM Patient Registry (https://www.dm-registry.org/uk/) aims to recruit any individual, from anywhere within the United Kingdom, with a diagnosis of myotonic dystrophy. Participants may be referred to the registry by health care professionals, or genetic testing/laboratory centres who are aware of the registry. Alternatively, a participant may have discovered the registry via promotional activities or by their own online searches. After completing the consent process, participants are able to enter information on to the registry platform (note all forms are also available offline as well). This is an ongoing database and all participants will invited to update their information on an annual basis.

The registry is sponsored by Muscular Dystrophy UK, Cure-DM and the Myotonic Dystrophy Support Group.

The database is divided into two main sections:

1. Mandatory items (demographic information, clinical diagnosis, genetic test result, current best motor function and wheelchair use) and
2. Highly encouraged items (severity of muscle symptoms, cardiac status, respiratory function, digestion, cataracts, and fatigue, ethnic origin and data on involvement with other registries)

The database is designed to be self reporting, however where specialised clinical or genetic information is required, the neuromuscular specialist in charge of the participants care can be invited to provide some additional information. The participant is able to select a health care provider from a pre-populated list at registration stage, if they wish to (optional feature). This information is included in the patient information and consent.

ELIGIBILITY:
Inclusion Criteria:

* All patients with a confirmed Myotonic Dystrophy diagnosis (or pending diagnosis) are eligible for inclusion. Diagnosis will be confirmed via genetic testing results

Exclusion Criteria:

* There are no exclusion criteria for the registry

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with Myotonic Dystrophy will volunteer to participate in this study. The study will be advertised through neuromuscular disease clinics, the registry website, patient organisations and conferences and meetings throughout the UK.
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2013-05 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Patient questionnaire | 12 months
  Patient reported myotonic dystrophy clinical diagnosis, symptoms relating to muscle weakness, motor function, medication use, family history and ethnicity.
Clinician questionnaire | 12 months
  Clinician reported patient cardiac measures, medication use, respiratory measures and genetic confirmation of myotonic dystrophy.

CONTACTS AND LOCATIONS:
Overall Officials: Chiara Marini-Bettolo, MD, PhD, Principal Investigator — John Walton Muscular Dystrophy Research Centre
Locations (1):
- John Walton Muscular Dystrophy Research Centre, Newcastle upon Tyne, United Kingdom

REFERENCES:
- [Result] Wood L, Cordts I, Atalaia A, Marini-Bettolo C, Maddison P, Phillips M, Roberts M, Rogers M, Hammans S, Straub V, Petty R, Orrell R, Monckton DG, Nikolenko N, Jimenez-Moreno AC, Thompson R, Hilton-Jones D, Turner C, Lochmuller H. The UK Myotonic Dystrophy Patient Registry: facilitating and accelerating clinical research. J Neurol. 2017 May;264(5):979-988. doi: 10.1007/s00415-017-8483-2. Epub 2017 Apr 10. PMID 28397002
- [Result] Best AF, Hilbert JE, Wood L, Martens WB, Nikolenko N, Marini-Bettolo C, Lochmuller H, Rosenberg PS, Moxley RT 3rd, Greene MH, Gadalla SM. Survival patterns and cancer determinants in families with myotonic dystrophy type 1. Eur J Neurol. 2019 Jan;26(1):58-65. doi: 10.1111/ene.13763. Epub 2018 Sep 16. PMID 30051542
- [Result] Alsaggaf R, Wang Y, Marini-Bettolo C, Wood L, Nikolenko N, Lochmuller H, Greene MH, Gadalla SM. Benign and malignant tumors in the UK myotonic dystrophy patient registry. Muscle Nerve. 2018 Feb;57(2):316-320. doi: 10.1002/mus.25736. Epub 2017 Jul 24. PMID 28662292
- [Result] Wood L, Bassez G, Bleyenheuft C, Campbell C, Cossette L, Jimenez-Moreno AC, Dai Y, Dawkins H, Manera JAD, Dogan C, El Sherif R, Fossati B, Graham C, Hilbert J, Kastreva K, Kimura E, Korngut L, Kostera-Pruszczyk A, Lindberg C, Lindvall B, Luebbe E, Lusakowska A, Mazanec R, Meola G, Orlando L, Takahashi MP, Peric S, Puymirat J, Rakocevic-Stojanovic V, Rodrigues M, Roxburgh R, Schoser B, Segovia S, Shatillo A, Thiele S, Tournev I, van Engelen B, Vohanka S, Lochmuller H. Eight years after an international workshop on myotonic dystrophy patient registries: case study of a global collaboration for a rare disease. Orphanet J Rare Dis. 2018 Sep 5;13(1):155. doi: 10.1186/s13023-018-0889-0. PMID 30185236